CLINICAL TRIAL: NCT01214759
Title: A Pilot Project to Assess the Safety and Tolerability of Truvada Plus Raltegravir as Post-exposure Prophylaxis (nPEP) Following Sexual Exposure to Human Immunodeficiency Virus (HIV)
Brief Title: Truvada Plus Raltegravir for Nonoccupational Post-exposure Prophylaxis (nPEP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Karen Vigil, Assistant Professor - Internal Medicine, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UT-NPEP
Record Dates: First submitted 2010-09-30; First posted 2010-10-05 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: HIV
Keywords: HIV; prevention; prophylaxis; Raltegravir; Truvada
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Truvada and Raltegravir (Other): Single arm
  Interventions: Drug: Truvada; Drug: Raltegravir

INTERVENTIONS:
Drug: Truvada — Tenofovir 200mg/emtricitabine 300mg once a day
  Other Names: Tenofovir 200mg/emtricitabine 300mg
Drug: Raltegravir — Raltegravir 400mg twice a day
  Other Names: Isentress

SUMMARY:
This study will evaluate the safety and tolerability of the combination of truvada and raltegravir given for 28 days for the prevention of HIV infection.

DETAILED DESCRIPTION:
Non-Occupational Post-Exposure Prophylaxis (nPEP) after sexual exposure to HIV is recommended by the Centers for Disease Control (CDC). Although no efficacy data exist for Post-Exposure Prophylaxis (PEP) after sexual exposure, PEP has been shown to reduce HIV transmission in other exposure situations such as occupational exposures and mother-to-child transmission. The role in nPEP of the newer agents approved for the treatment of HIV infection remains unknown. The anti-HIV drug raltegravir works early in the life cycle of the virus, before it integrates with human DNA. It has few side effects and drug interactions what makes it an ideal drug for an nPEP regimen.

We aim to asses the safety and tolerability of the combination of truvada and raltegravir for nPEP.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* HIV uninfected on the basis of a negative HIV rapid test, EIA or Western blot, and without any signs or symptoms of acute HIV infection
* Able to understand and provide consent
* High-Risk Exposure Characteristic (One or more of the below, unprotected or with failed condom use):

  * Receptive Anal Intercourse
  * Insertive Anal Intercourse
  * Receptive Vaginal Intercourse
  * Insertive Vaginal Intercourse
  * Receptive Oral Intercourse with Intraoral Ejaculation with known HIV+ source
* High-Risk Source (One or more of the below):

  * Known HIV positive
  * MSM
  * MSM/W
  * CSW
* Sexual perpetrator Partner of one of the above
* Exposure within 72 hours of presentation
* Not known to be HIV-1 positive
* No countermanding concomitant medications or allergies

Exclusion Criteria:

* Patients <18 years of age
* Unable to understand and provide consent
* Non-occupational exposure to HIV-1 not recent enough to commence the first dose of study medication within 72 hours from the exposure
* Known to be HIV positive
* Any condition which in the opinion of the intake provider will seriously compromise the patient's ability to comply with the protocol, including adherence to nPEP medication
* Demonstrated HIV-1 positive on rapid testing
* Unwillingness to commit to barrier-method (male and/or female condom) use until HIV negative status is confirmed 6 months after exposure
* Unwillingness of breast-feeding women to transition to formula feeding
* Any active psychiatric illness or active drug or alcohol abuse that, in the opinion of the investigator, could prevent compliance with study procedures
* Pregnancy
* Chronic hepatitis B infection, diagnosed by either positive serum HBsAg or positive serum HBV DNA; or prior lamivudine or other therapy for hepatitis B
* Creatinine clearance less than 30 mL/min as calculated by Cockcroft-Gault formula
* Unwillingness to participate in study procedures, including Mental Health referral and intervention
* Known intolerance or allergy to tenofovir DF, emtricitabine or raltegravir
* Use of prohibited concomitant medication: dilantin, phenobarbital and rifampin which cannot be used with raltegravir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Vigil, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Smith DK, Grohskopf LA, Black RJ, Auerbach JD, Veronese F, Struble KA, Cheever L, Johnson M, Paxton LA, Onorato IM, Greenberg AE; U.S. Department of Health and Human Services. Antiretroviral postexposure prophylaxis after sexual, injection-drug use, or other nonoccupational exposure to HIV in the United States: recommendations from the U.S. Department of Health and Human Services. MMWR Recomm Rep. 2005 Jan 21;54(RR-2):1-20. PMID 15660015
- [Background] Pinkerton SD, Martin JN, Roland ME, Katz MH, Coates TJ, Kahn JO. Cost-effectiveness of HIV postexposure prophylaxis following sexual or injection drug exposure in 96 metropolitan areas in the United States. AIDS. 2004 Oct 21;18(15):2065-73. doi: 10.1097/00002030-200410210-00011. PMID 15577628
- [Background] Kahn JO, Martin JN, Roland ME, Bamberger JD, Chesney M, Chambers D, Franses K, Coates TJ, Katz MH. Feasibility of postexposure prophylaxis (PEP) against human immunodeficiency virus infection after sexual or injection drug use exposure: the San Francisco PEP Study. J Infect Dis. 2001 Mar 1;183(5):707-14. doi: 10.1086/318829. Epub 2001 Feb 1. PMID 11181146
- [Background] Tsai CC, Follis KE, Sabo A, Beck TW, Grant RF, Bischofberger N, Benveniste RE, Black R. Prevention of SIV infection in macaques by (R)-9-(2-phosphonylmethoxypropyl)adenine. Science. 1995 Nov 17;270(5239):1197-9. doi: 10.1126/science.270.5239.1197. PMID 7502044

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Truvada and Raltegravir
Started | 103
28 Days nPEP Completion | 85
Completed | 55
Not Completed | 48

BASELINE CHARACTERISTICS:
Population: All who were enrolled
Arm/Group | Truvada and Raltegravir
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 92
Region of Enrollment [Number; unit: participants]
  United States | 103

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Assessed by the Number of Participants Who Were HIV Positive at 6 Months
Description: This measure assesses whether the combination of Truvada and Raltegravir prevents the acquisition of HIV at six months among HIV-negative people who have been exposed to HIV.
Time Frame: 6 months
Population: All who completed all study visits
Measure: Number; unit: participants
Arm/Group | Truvada and Raltegravir
Number analyzed (Participants) | 55
participants | 0

2. Secondary Outcome: Number of Participants Exhibiting Clinical or Laboratory Abnormalities Resulting From the 28-day Exposure to the Antiretroviral Drugs Being Explored in This Study
Description: Participants who experienced side effects categorized as grade 3 or higher by the Division of AIDS table for grading the severity of adult and pediatric adverse events were tested for clinical or laboratory abnormalities.
Time Frame: 28 days
Population: Only participants who experienced side effects categorized as grade 3 or higher by the Division of AIDS table were tested for clinical or laboratory abnormalities, and since no participants experienced side effects greater than grade 1, no participants were tested for clinical or laboratory abnormalities.
Arm/Group | Truvada and Raltegravir
Number analyzed (Participants) | 0

3. Secondary Outcome: Safety and Tolerability as Assessed by the Number of Participants Who Completed the 28-day Course of the Antiretroviral Drugs Being Explored in This Study
Time Frame: 28 days
Population: All who were enrolled
Measure: Number; unit: participants
Arm/Group | Truvada and Raltegravir
Number analyzed (Participants) | 103
participants | 85

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed at follow up visits at 2 weeks, 4 weeks, 3 months, and 6 months.
Description: All adverse events that occurred are categorized as grade 1 (mild) by the Division of AIDS table for grading the severity of adult and pediatric adverse events. No grade 2 (moderate), grade 3 (severe), or grade 4 (potentially life threatening) adverse events occurred.
Arm/Group | Truvada and Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 8/85
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Truvada and Raltegravir (N=85)
Headache (General disorders) | 6 (6)
Fatigue (General disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (4)
Dizziness (General disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Flushing (General disorders) | 2 (2)
Loose stools (Gastrointestinal disorders) | 2 (2)
Delayed menstruation (Reproductive system and breast disorders) | 1 (1)
Decreased appetite (General disorders) | 1 (1)
Nightmares (General disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Face pain (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a pilot study with a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes